CLINICAL TRIAL: NCT05809817
Title: Economic Evaluation of the Current Proposal and Different Decision-making Scenarios of Coverage Increases of an Oral Health Policy for Patients With Type 2 Diabetes Mellitus in Chile: A Microsimulation Model Based on Real-world Data
Brief Title: Oral Health Policy for Patients With Type 2 Diabetes Mellitus in Chile: A Microsimulation Model Based on Real-world Data
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Chile (Other)
Responsible Party: Sponsor
Other Study IDs: FONIS SAI0060
Record Dates: First submitted 2023-03-10; First posted 2023-04-12 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-03

CONDITIONS: Type 2 Diabetes Mellitus; Periodontitis; Diabetic Complication; Dental Care
Keywords: Periodontics; Periodontal Medicine; Type 2 Diabetes Mellitus; Non-surgical Periodontal Therapy; Diabetic complication; Cost-Effectiveness Analysis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Periodontitis; Diabetes Complications | interventions — Periodontal Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention (Periodontal treatment): Patients with T2DM under follow-up in the PSCV will receive the usual periodontal therapy performed at the CEMO Villa Sur in the commune of Pedro Aguirre Cerda and at the CESFAM Puerto Varas in the context of PSCV. The care protocols and national evidence establish that the standard treatment of periodontitis consists of 4 or more sessions of scaling and root planing per sextant, depending on the severity of the disease.
  Interventions: Procedure: Periodontal treatment
- Control (Matched, non-active intervention): Patients with T2DM under follow-up in the PSCV, with non-active control (withouth periodontal treatment) that will be matched in a ratio of 1:1 through Propensity Score Matching according to baseline HbA1c levels and demographic baseline data (age, sex).

INTERVENTIONS:
Procedure: Periodontal treatment — Scaling and root planing
  Groups: Intervention (Periodontal treatment)

SUMMARY:
The goal of this study is to evaluate the cost-effectiveness of the current proposal and different decision-making scenarios of periodontal care coverage increases for patients with T2DM in Chile. The main objective of the clinical section of this study (effectiveness) aims to determine the effectiveness of periodontal care in patients with T2DM under follow-up in the Cardiovascular Health Program (Programa de Salud Cardiovascular, PSCV) of the in the CEMO Villa Sur of Pedro Aguirre Cerda and the CESFAM Antonio Varas of Puerto Montt.

A highly matched control group is proposed using Propensity Score Matching of PSCV patients with T2DM who have not received periodontal care. This would allow a better comparison of the individuals who will actually be treated against a counterfactual against of those with similar characteristics who did not receive periodontal intervention during the follow-up period of this first stage.

DETAILED DESCRIPTION:
Introduction: Oral diseases and type 2 Diabetes Mellitus (T2DM) constitute an important public health problem in Chile, due to their high prevalence and economic and social impact. T2DM increases the risk of oral diseases such as periodontitis, and the latter worsens the metabolic control of T2DM, increasing the risk of macrovascular and microvascular complications. More than 10% of total health spending in Chile is allocated to the treatment of T2DM, especially for the management of its complications. The main T2DM control program in Chile is the Cardiovascular Health Program (PSCV) that treats more than 900,000 people with T2DM, however, its results are still insufficient. Although periodontal treatment improves the metabolic control of T2DM, the proposed goal of periodontal care coverage for patients with T2DM in the context of the PSCV is only 2%. Therefore, the decision to expand periodontal care coverage to efficiently improve the health status of these patients is crucial.

Objective: To evaluate the cost-effectiveness of the current proposal and different decision-making scenarios for increasing periodontal care coverage for patients with T2DM from the perspective of the public health system in Chile.

Methods: In the first stage, a prospective observational cohort study will be conducted at the CEMO Villa Sur in Pedro Aguirre Cerda and at the CESFAM Puerto Varas in the commune of Puerto Montt to estimate treatment costs and the effectiveness of periodontal care on glycated hemoglobin (HbA1c) levels in the context of PSCV (real-world data). The intervention cohort will consist of those patients with T2DM receiving periodontal care during 2023, while the comparison cohort will consist of those on the waiting list during the same period, matched 1:1 through Propensity Score Matching. In a second stage the costs and effects of each coverage alternative (2%, 20%, 40%, 60%, 80% and 100%) will be modeled using microsimulation techniques to estimate the projected impact over a lifetime horizon of HbA1c changes on the risk of complications, death and decreased quality of life. Costs for each clinical stage will be obtained from national GES (Explicit Health Guarantees) cost estimates, supplemented by other sources, and quality-adjusted life years will be used as a summary measure of effects. Costs and effects will be combined to estimate the incremental cost-effectiveness ratio (ICER). From the probabilistic sensitivity analysis, acceptability curves and frontiers and expected loss curves for the proposed courses of action will be estimated.

ELIGIBILITY:
* Inclusion criteria:

  1. Intervention: Patients with T2DM under follow-up in the PSCV who present records of HbA1c levels for the last three months prior to care and who receive complete periodontal treatment at the CEMO Villa Sur in the commune of Pedro Aguirre Cerda and at the CESFAM Puerto Varas in Puerto Montt under the PSCV will be selected.
  2. Control: A control cohort of patients with T2DM under follow-up in the PSCV will be determined, matching 1:1 through Propensity Score Matching according to baseline HbA1c levels and demographic baseline data (age and sex).
* Exclusion criteria:

  1. Patients with a history of periodontal treatment.
  2. Pregnant or breastfeeding.
  3. Time spent in PSCV<1year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with T2DM under follow-up in the PSCV
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Metabolic control | Baseline and 3 months after periodontal treatment
  Mean change from baseline HbA1c at 3 months after periodontal treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Baeza, DDS,MSc,PhD, Study Chair — Department of Conservative Dentistry, Faculty of Dentistry, University of Chile
Locations (2):
- Chile (2):
  - CESFAM Puerto VARAS, Puerto Varas, De Los Rios
  - CEMO Villa Sur, Santiago

IPD SHARING:
Plan to Share IPD: Undecided
The datasets generated during and/or analysed during the study will be available from the corresponding author on reasonable request.